CLINICAL TRIAL: NCT03101891
Title: Renal Anhydramnios Fetal Therapy (RAFT) Trial
Brief Title: Renal Anhydramnios Fetal Therapy
Acronym: RAFT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00164021; R01HD100540 (NIH)
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Anhydramnios; Potter Syndrome; Lung Hypoplasia; Multicystic Dysplastic Kidney; Multicystic Renal Dysplasia, Bilateral; Lower Urinary Tract Obstructive Syndrome; Fetal Renal Anomaly
Keywords: Amnioinfusion; Fetal therapy; Bilateral Renal Agenesis; Fetal Renal Failure; Lower Urinary Tract Obstruction (LUTO); Anhydramnios
MeSH Terms: conditions — Hereditary renal agenesis; Multicystic Dysplastic Kidney; Multicystic renal dysplasia, bilateral | interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: All eligible patients will be offered participation in the study. Participants can elect for invasive therapy with amnioinfusions or expectant management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Serial amnioinfusions with isotonic fluid (Experimental): There are two interventional arms to the trial. Recruitment in the bilateral renal agenesis arm of the trial was stopped in July 2022 after Data Safety Monitoring Board (DSMB) review.
  Recruitment is ongoing in the non-bilateral renal agenesis, fetal renal failure with anhydramnios arm of the trial. Patients will undergo amnioinfusions with isotonic fluid every 2-12 days.. A spinal needle will be used to perform the infusion. The latest infusions will begin is 26 weeks gestation. Standard postnatal care will occur at a RAFT center.
  Interventions: Procedure: Serial amnioinfusions with isotonic fluid; Device: Spinal needle; Drug: Isotonic fluid
- Expectant (No Intervention): Patients will be observed serially by ultrasound, fetal echocardiogram and MRI. Standard postnatal care will occur at a RAFT center.

INTERVENTIONS:
Procedure: Serial amnioinfusions with isotonic fluid — Amnioinfusions will be performed by an expert in fetal procedures with a 20 or 22 gauge needle using sterile technique and ultrasound guidance. Local anesthetic will be employed. The fluid will consist of warmed isotonic fluid. Infusions may take up to 1 hour.
  Other Names: Renal Anhydramnios Fetal Therapy (RAFT)
  Arms: Serial amnioinfusions with isotonic fluid
Device: Spinal needle — A 20 or 22 gauge spinal needle will be used with sterile technique to access the uterus under ultrasound guidance and to infuse isotonic fluid.
  Other Names: Obstetrics and gynecology needle
  Arms: Serial amnioinfusions with isotonic fluid
Drug: Isotonic fluid — Isotonic fluids, including normal saline or lactated ringers solution, will be infused into the uterus through a spinal needle under ultrasound guidance using sterile technique. This fluid will act as replacement amniotic fluid.
  Other Names: Normal saline; Lactated ringers solution
  Arms: Serial amnioinfusions with isotonic fluid

SUMMARY:
Early pregnancy renal anhydramnios (EPRA) is a condition where a pregnant woman does not have any amniotic fluid around her fetus because of a problem with the fetus's kidneys. This condition is thought to be fatal once the fetus is born because of inadequate lung growth. The Renal Anhydramnios Fetal Therapy (RAFT) Trial offers eligible pregnant women with a diagnosis of EPRA an experimental therapy of repeated or serial "amnioinfusions" of fluid into the womb. An amnioinfusion involves placing a small needle through the pregnant woman's skin into the womb next to the fetus. Warm sterile fluid with balanced electrolytes and antibiotics is then slowly infused into amniotic space inside the womb. The aim is to help the fetus's lungs grow enough so he or she can survive after birth. These amnioinfusions will be carried out by an expert in fetal interventions at a RAFT center. There is a significant risk of early rupture of membranes and early delivery in subjects who receive amnioinfusions, and any potential trial participants will be counseled about these risks before they decide whether to join the trial. Any eligible patients who, after counseling, elect to terminate the pregnancy will not be eligible to participate in the trial. All eligible patients who choose to join the RAFT trial will be able to choose their assignment into one of two arms of the study: (1) to receive serial amnioinfusions (2) to not receive amnioinfusions but receive monitoring for the remainder of the pregnancy at the RAFT center. Thus, assignment of patients to study arm will not be random, but will be decided by the participant. Fetuses who do survive after birth will require intensive medical management for kidney failure including placement of a dialysis catheter and dialysis therapy with the eventual need for a kidney transplant. Treatment for lung disease secondary to abnormal lung development may also be required. The study will follow babies and their families until non-survival or transplant.

Update: Due to recommendations from the RAFT trial Data and Safety Monitoring Board, the trial is no longer open to enrollment for pregnancies complicated by bilateral renal agenesis as of July 19, 2022. Enrollment for patients with pregnancies complicated by other causes of fetal renal failure remains open.

DETAILED DESCRIPTION:
Amniotic fluid is critical for normal lung development. After the first trimester of pregnancy amniotic fluid is composed nearly completely of fetal urine. The absence of amniotic fluid due to lack of urine production by the fetal kidneys is known as anhydramnios. Early pregnancy renal anhydramnios or EPRA is thought to be 100% lethal after birth if left untreated because of neonatal respiratory failure. The two causes of EPRA are bilateral renal agenesis or fetal renal failure (such as from multicystic dysplastic kidneys or obstructed kidneys). Recently there have been clinical case reports of repeated or serial infusions of isotonic fluid (amnioinfusions) into the amniotic cavity leading to respiratory survival in neonates with a history of EPRA. Some surviving neonates have gone on to undergo successful dialysis and kidney transplant as toddlers. However, no prospective trial has investigated the safety of amnioinfusions in EPRA, the feasibility of doing serial amnioinfusions in EPRA pregnancies without causing rupture of membranes, or the neonatal survival rate after serial amnioinfusions for EPRA. Accordingly the goal of the Renal Anhydramnios Fetal Therapy (RAFT) trial is to determine the safety, feasibility, and efficacy of serial amnioinfusions to promote normal fetal lung development in EPRA. Pregnant patients presenting to a RAFT center with a diagnosis of EPRA will undergo an evaluation including diagnostic amnioinfusion with ultrasound imaging to verify the diagnosis. Counseling by a team of subspecialists including a maternal fetal medicine doctor, a pediatric nephrologist, a pediatric surgeon, a neonatologist, a kidney transplant specialist, a genetic counselor and a social worker will be given to every patient. This counseling is meant to provide the clearest picture possible of what serial amnioinfusions entail and what life will be like for a surviving neonate with no kidney function. Survivors will require urgent dialysis with a peritoneal or hemodialysis catheter. These children are prone to significant infections and often need a gastrostomy tube in order to receive sufficient nutrition. The goal is for these children to ultimately undergo the most robust form of renal replacement therapy with a kidney transplant once they are large enough to tolerate it.

Once the diagnosis of EPRA is confirmed, counseling is complete and a patient is deemed eligible for serial amnioinfusions, enrollment into the study will be offered. Patients may choose to enroll in the study, may choose to continue the pregnancy and not be a part of the study or may choose to terminate the pregnancy. If the patients elect to enroll in the study, they will be given a further choice of intervention with serial amnioinfusions or expectant management with repeat imaging. Participants will not be randomized because there is no realistic hope that expectant management will lead to postnatal survival. Patients who do not choose to undergo amnioinfusions but who also do not elect to terminate will provide invaluable insight into the in utero natural history of EPRA if they enroll in the trial. The sample size of this trial is based on a calculation of the number of patients required to adequately determine a postnatal survival rate of amnioinfusions for EPRA with narrow confidence intervals. Postnatal survival will be defined as survival for >=14 days and placement of dialysis access; this is the primary outcome measure. We have determined that 35 maternal/fetal participants are required in order to calculate a survival rate of anywhere from 20-80%. We plan to study two 35 participant cohorts of EPRA patients, those with EPRA from bilateral renal agenesis and those with EPRA from fetal renal failure. We will therefore aim for a total of 70 maternal/fetal pairs with EPRA to undergo serial amnioinfusions. Additionally we will aim to recruit 30 maternal/fetal pairs with EPRA in the expectant management group for a total of 100 participants.

During the prenatal portion of the trial we plan to collect a small specimen of amniotic fluid from participants in the amnioinfusion group during each amnioinfusion. This fluid will be assayed for different protein and lipid measures of lung maturity at a research lab at Johns Hopkins. Additionally, in both the amnioinfusion group and the expectant management group we will study ultrasound, MRI and echocardiogram measures of lung growth. We will correlate these biochemical and radiologic markers with survival in order to better understand who is likely to respond to amnioinfusions and why that response is occurring. We also plan to study several secondary and tertiary outcomes in our surviving EPRA patients. These outcomes include survival to discharge from a RAFT center, survival to transplant and quality of life measures for both participants and their families.

The changes made to the outcomes are due to the protocol amendment.

Update: Due to recommendations from the RAFT trial Data and Safety Monitoring Board, the trial is no longer open to enrollment for pregnancies complicated by bilateral renal agenesis as of July 19, 2022. Enrollment for patients with pregnancies complicated by other causes of fetal renal failure remains open.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed anhydramnios before 22 weeks gestational age (GA) for patients with fetal renal failure (excluding bilateral renal agenesis)
2. Consent is signed and first therapeutic amnioinfusion can and does occur before 26 weeks and 0 days GA
3. Confirmation that the expectant mother does not wish to undergo termination of the pregnancy
4. Age ≥ 18 years of age for expectant mothers
5. Willingness to be followed and deliver at a RAFT center
6. Willingness for postnatal care to be performed at a RAFT center until discharge
7. Completed consults with Pediatric Nephrology, Neonatology, Transplant Surgery, Pediatric surgery, Maternal-Fetal Medicine Specialist, and Licensed Clinical Social Worker and a Genetic Counselor

Exclusion Criteria:

1. Cervix less than 2.5 cm in length
2. No significant pathogenic or likely significant pathogenic findings on Karyotype or Microarray
3. Other significant congenital anomalies in the fetus
4. Evidence of chorioamnionitis or abruptio placentae
5. Evidence of rupture of membranes or chorioamniotic separation
6. Evidence of preterm labor
7. Multiple gestation
8. Severe maternal medical condition in pregnancy.
9. Maternal depression as assessed by a Beck Depression Inventory score equal to or greater than 17 that is refractory to treatment
10. Technical limitations precluding amnioinfusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women are the focus of this study
Enrollment: 70 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of neonates surviving to >= 14 days and placement of dialysis access after serial amnioinfusions | Birth to either survival to >=14 days and placement of dialysis access, or nonsurvival, up to 3 weeks
  The proportion of neonates who survive to >= 14 days and placement of dialysis access as well as the exact confidence interval will be presented for CoBRA and fetal renal failure (FRF) patients separately in the intervention group.

SECONDARY OUTCOMES:
Number of infusions before rupture of membrane among those in the intervention arm | During the EPRA pregnancy, up to 9 months
  The feasibility of serial amnioinfusions for EPRA will be measured the number of infusions prior to rupture of membrane among those in the intervention arm
Mean gestational age at the time of rupture of membrane among those in the intervention arm | During the EPRA pregnancy, up to 9 months
  The feasibility of serial amnioinfusions for EPRA will be measured using the mean gestational age at rupture among those in the intervention arm
Mean gestational age at delivery among those in the intervention arm | During the EPRA pregnancy, up to 9 months
  The feasibility of serial amnioinfusions for EPRA will be measured using the mean gestational age at delivery among those in the intervention arm
Rate of in utero fetal demise among those in the non-intervention arm | During the EPRA pregnancy, up to 9 months
  We will perform an exploratory study of the in utero natural history of untreated EPRA by examining the rate of in utero fetal demise among those in the non-intervention arm.
Mean gestational age at delivery among those in the non-intervention arm | During the EPRA pregnancy, up to 9 months
  We will perform an exploratory study of the in utero natural history of untreated EPRA by examining the mean gestational age among those in the non-intervention arm
Correlations between fetal ultrasound, echocardiogram MRI biomarkers as well as amniotic fluid biomarkers, and the success of RAFT for EPRA | End of follow-up, up to 4 years after transplant
  The correlations between fetal ultrasound, echocardiogram MRI biomarkers as well as amniotic fluid biomarkers and the success of RAFT for EPRA will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Atkinson, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (9):
  - University of Southern California/Children's Hospital of Los Angeles/Huntington Hospital, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Hare EM, Jelin AC, Miller JL, Ruano R, Atkinson MA, Baschat AA, Jelin EB. Amnioinfusions to Treat Early Onset Anhydramnios Caused by Renal Anomalies: Background and Rationale for the Renal Anhydramnios Fetal Therapy Trial. Fetal Diagn Ther. 2019;45(6):365-372. doi: 10.1159/000497472. Epub 2019 Mar 21. PMID 30897573
- [Background] Huber C, Shazly SA, Blumenfeld YJ, Jelin E, Ruano R. Update on the Prenatal Diagnosis and Outcomes of Fetal Bilateral Renal Agenesis. Obstet Gynecol Surv. 2019 May;74(5):298-302. doi: 10.1097/OGX.0000000000000670. PMID 31098643
- [Result] Bienstock JL, Birsner ML, Coleman F, Hueppchen NA. Successful in utero intervention for bilateral renal agenesis. Obstet Gynecol. 2014 Aug;124(2 Pt 2 Suppl 1):413-415. doi: 10.1097/AOG.0000000000000339. PMID 25004316
- [Derived] Miller JL, Baschat AA, Rosner M, Blumenfeld YJ, Moldenhauer JS, Johnson A, Schenone MH, Zaretsky MV, Chmait RH, Gonzalez JM, Miller RS, Moon-Grady AJ, Bendel-Stenzel E, Keiser AM, Avadhani R, Jelin AC, Davis JM, Warren DS, Hanley DF, Watkins JA, Samuels J, Sugarman J, Atkinson MA. Neonatal Survival After Serial Amnioinfusions for Bilateral Renal Agenesis: The Renal Anhydramnios Fetal Therapy Trial. JAMA. 2023 Dec 5;330(21):2096-2105. doi: 10.1001/jama.2023.21153. PMID 38051327
- [Derived] Atkinson MA, Jelin EB, Baschat A, Blumenfeld YJ, Chmait RH, O'Hare E, Moldenhauer JS, Zaretsky MV, Miller RS, Ruano R, Gonzalez JM, Johnson A, Mould WA, Davis JM, Hanley DF, Keiser AM, Rosner M, Miller JL. Design and Protocol of the Renal Anhydramnios Fetal Therapy (RAFT) Trial. Clin Ther. 2022 Aug;44(8):1161-1171. doi: 10.1016/j.clinthera.2022.07.001. Epub 2022 Jul 30. PMID 35918190
- See also: The Center for Fetal Therapy — http://www.hopkinsmedicine.org/gynecology_obstetrics/specialty_areas/fetal_therapy/